CLINICAL TRIAL: NCT03843983
Title: Lipiflow Effect on Lacrimal Meibum Composition and on Adverse Environmental Conditions in Subjects With Meibomian Gland Dysfunction
Brief Title: Effect of Thermal Pulsation System (Lipiflow) Treatment for Ocular Surface Disease Due to Meibomian Gland Dysfunction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Instituto Universitario de Oftalmobiología Aplicada (Institute of Applied Ophthalmobiology) - IOBA (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IOBA-2019-2
Record Dates: First submitted 2019-02-05; First posted 2019-02-18 (Actual); Last update posted 2021-06-03 (Actual); Status verified 2021-05

CONDITIONS: Evaporative Dry Eye Disease
Keywords: Meibomian gland dysfunction; Lipiflow; Meibum composition; Adverse environmental conditions; Dry eye disease
MeSH Terms: conditions — Dry Eye Syndromes; Meibomian Gland Dysfunction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Lipiflow treatment (Other): Lipiflow® application: Treated with Lipiflow. All patients in this study are treated with Lipiflow once.
  Interventions: Device: Lipiflow® application

INTERVENTIONS:
Device: Lipiflow® application — Lipiflow® will be applicated in both lids of each eye during 12 minutes once. Firstly, a drop of anesthetic will be instilled in each eye. Then, while the participant stays with his eyes closed, a one-used applicator will be placed covering the subject's lid. The instrument applies heat and pressure in the lid during 12 minutes. Time frame: between 2 and 7 days after visit 1.
  Then, there will be 3 follow-up visits in 3, 6 and 12 months after treatment.

SUMMARY:
Meibomian glands are a kind of sebaceous gland located in the tarsus of lower and upper lids and their function is to express lipids to the tear film. The secretion of lipids, polar and no-polar, produced in the Meibomian glands is denominated as meibum and it forms the external layer of the tear film. Its thickness varies from 15 to 200 nm and it is related with the tear film stability and the evaporation of the tear film.

The meibum composition is variable among participants, especially in those who suffer Meibomian gland dysfunction or dry eye disease. Meibomian gland dysfunction is the leading cause of ocular surface disease.

Meibomian gland dysfunction management depends on its severity, but eyelid hygiene, including warming and expression of Meibomian gland, is recommended from clinical stage 1 and it has proven its efficacy. However, lack of participant compliance can be a problem when this therapy is prescribed. In the last few years, some devices have been developed to improve the efficacy of this therapy, as for example the application of Vectored Thermal Pulsation with the Lipiflow device.

It has been reported that low relative humidity values increase evaporative rates in both dry eye participants and healthy participants. Also, our group has extensively proven the negative effect of adverse environments (in the Controlled Environment Laboratory (CELab)) in clinical variables such as tear stability, dry eye symptoms and corneal staining both in healthy and dry eye participants.

Therefore, the hypothesis of this study is that improving the Meibomian gland secretion through the application of warm and pressure with Lipiflow device, meibum composition would change in participants with Meibomian gland dysfunction and they would be less affected by adverse environmental conditions simulated in a controlled environmental chamber.

The study will try to assess the effect of Lipiflow on the meibum in patients exposed to controlled adverse environmental conditions.

DETAILED DESCRIPTION:
Justification:

Meibomian glands are a kind of sebaceous gland located in the tarsus of lower and upper lids and their function is to express lipids to the tear film. Each gland consists of several acini surrounding a central conduct and connected to it by conducts. The internal side f the gland is not visible, while the external one is located in the lid margin, before the muco-cutaneous junction, where they express the lipids to the tear film. Meibomian glands from lower lids are thicker than those of upper lid.

The secretion of lipids, polar and no-polar, produced in the Meibomian glands is denominated as meibum and it forms the external layer of the tear film. Its thickness varies from 15 to 200 nm and it is related with the tear film stability and the evaporation of the tear film. The lipid layer is divided in two sub-layers: the no-polar external part and the polar internal part. This internal part creates and inter-phase between the tear film muco-aqueous layer and the lipid no-polar layer, contributing to its stability. The no-polar lipids retards the evaporation of the aqueous component of the tear film so, inhibits the inflammation produced by the evaporation.

The meibum composition is variable among participants, especially in those who suffer meibomian gland dysfunction or dry eye disease.

Meibomian Gland Dysfunction is the leading cause of ocular surface disease. There has been substantial confusion regarding its definition and the origin of its symptoms. In part because of this uncertainty, the prevalence of this disease is unknown, and numbers are highly variable. A survey performed in the USA estimated a prevalence of 37 percentage and 47 percentage as reported by ophthalmologists and optometrists, respectively.

Meibomian gland dysfunction management depends on its severity, but eyelid hygiene, including warming and expression of Meibomian gland, is recommended from clinical stage 1 and it has proven its efficacy. However, lack of participant compliance can be a problem when this therapy is prescribed. In the last few years, some devices have been developed to improve the efficacy of this therapy, as for example the application of Vectored Thermal Pulsation with the Lipiflow device.

Lipiflow has proven its efficacy in the short term (3 months), however there is scarce information about its sustained effect in the long therm. To the best of our knowledge, there are only two long-term studies, where a positive effect in Meibomian glands function and dry eye symptoms has been reported after 12 months and 3 years of follow-up. People are constantly exposed to adverse environments, such as low humidity or presence of air flow, especially when are indoors (air-conditioned offices, transportation means…). It has been reported that low relative humidity values increase evaporative rates in both dry eye participants and healthy participants. Likewise, higher relative humidity increases tear break-up time (TBUT) values, a reflection of improved tear film stability, presumably through decreased evaporation. Also, our group has extensively proven the negative effect of adverse environments (in the Controlled Environment Laboratory (CELab)) in clinical variables such as tear stability, dry eye symptoms and corneal staining both in healthy and dry eye participants.

Hypothesis:

By improving the Meibomian gland secretion through the application of heat and pressure with Lipiflow device, meibum composition would change in participants with Meibomian gland dysfunction and they would be less affected by adverse environmental conditions simulated in a controlled environmental chamber.

Objective:

To evaluate the effect of Lipiflow application on the meibum composition and if there is a variation on symptoms and sings in participants with ocular surface disease due to Meibomian gland dysfunction who are exposed to adverse environmental conditions.

Study plan:

Participants will perform a total of 10 visits (in 6 days): an inclusion visit (V0), two basal visits (V1a, V1b), one treatment visit (V2) and six follow-up visits: at 3 (V3a, V3b), 6 (V4a, V4b) and 12 months (V5a, V5b) after treatment, respectively. Data from V0 and post treatment visits (V3-V5) will be compared and statistically evaluated.

V0: Recruitment visit. Participants attending the Ocular Immunology Unit (IOBA) with ocular surface disease due to Meibomian gland dysfunction will be recruited after checking inclusion and exclusion criteria. If eligible, participants will sign the informed consent and will be scheduled for V1 within the next 14 days.

V1: Baseline visit (V1a - V1b). Participants will come to the clinic without any artificial tear use four hours before the visit. Participants will enter the environmental chamber at CELab, where they will be exposed for 30 minutes to a normal controlled environment which consists of 23 degrees Celsius and 50 percentage relative humidity; then, tests will be performed still under normal controlled environment (Visit 1a).

Then, participants will be exposed for 2 hours to an adverse controlled environment consisting of 23 degrees Celsius and 10 percentage relative humidity, and the same tests as above will be performed (Visit 1b).

Between 2-7 days after, they will be scheduled for the next visit. V2: Treatment Visit. Participants will come to the clinic without any artificial tear use four hours before the visit. Lipiflow treatment will be applied following the manufacturer protocol.

V3-V5 (a and b): 3, 6- and 12-months post-treatment evaluations. Participants will come to the clinic without any artificial tear use four hours before the visit. Participants will be evaluated after 30 minutes of exposure to normal controlled environment in CELab. Right after, participants will be exposed to a 2 hours of adverse controlled environment exposure and the same tests as before will be performed.

Clinical evaluation and take of samples:

* Ocular symptoms questionnaires.
* Visual Acuity measure.
* Lid margin evaluation.
* Meibomian gland evaluation.
* Lid layer thickness measure (interferometry).
* Conjunctiva hyperemia evaluation.
* Non Invasive Break Up Time (NIBUT).
* Tear Break Up Time with fluorescein (TBUT).
* Corneal staining with fluorescein.
* Conjunctiva staining with lissamine green.
* Meibomian gland morphology evaluation (meibography).
* Collection and analysis of meibum samples.
* Lipiflow application.

Data Analysis:

Mean values and 95 percentage confidence intervals (95 percentage CI) will be used to describe quantitative variables, while median values and interquartile range will be used for ordinal ones. For primary efficacy endpoint, TBUT comparisons between V1a and V3a will be performed by t-Student test for two paired samples.

In addition, a linear mixed effects model will be used to evaluate the effect of time on clinical variables and Least Squares Means and their differences will be estimated for effect quantification. Tukey´s method will be used to compute the adjusted p-values for multiple comparisons. Ordinal scale variables will be modeled using cumulative logit ordinal models with a mixed-effect for evaluating changes over time.

ELIGIBILITY:
Inclusion Criteria:

* Age of 18 or older.
* Signature of informed consent form.
* Ocular Surface Index (OSDI) questionnaire score more or equal 13.
* Meibomian gland secretion score of the lower lid in both eyes less or equal 12 in the Meibomian Gland Yielding Liquid Secretion (MGYLS) Score.
* At least 10 out of 15 functioning MG of the lower eyelid, evaluated with the Meibomian Gland Evaluator (MGE).

Exclusion Criteria:

* Any ocular pathology other than Ocular Surface Disease due Meibomian Gland Dysfunction (MGD).
* Unwilling to abstain from the use of systemic or topical treatments for MGD or dry eye for the study duration (except for artificial tears, ocular lubricants or dietary supplements).
* Unwilling to abstain from the use of systemic medications known to cause dryness for the study duration.
* History of severe ocular inflammation or infection in the 6 previous months.
* Eyelid abnormalities that affect lid function.
* Any ocular surgery or trauma that may affect corneal sensitivity and/or normal tear distribution in the 6 previous months.
* Contact lens use must be stopped 15 days before inclusion and will not be resumed until the end of the study.
* Punctal plugs or punctal occlusion within the past three months.
* Pregnancy or breastfeeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2019-03-25 (Actual); Primary Completion 2020-10-13 (Actual); Study Completion 2020-10-13 (Actual)

PRIMARY OUTCOMES:
Tear break up time (TBUT) | 3 months after treatment
  Measure of tear film stability with fluorescein. Tear Break Up Time with fluorescein (TBUT): fluorescein sodium (Entod Research Cell United Kingdom Ltd, New Southgate, London, United Kingdom) will be instilled in the inferior conjunctiva. Tear film pattern will be observed through a slit lamp with blue light and yellow filter. Participants will be asked to blink three times and then maintain their eye open as longer as possible. The time between the last blink and the moment when the first black spot appears will be noted in seconds. This measure will be repeated three times and the average of them will be calculated. Measures lower than 8 seconds are considered no normal.

SECONDARY OUTCOMES:
Meibomian Gland Score (MGS) 12 months after treatment | 12 months after treatment
  Meibomian Gland Evaluator device will be used. This instrument applies a constant pressure of 1.25g/gmm^2 in 8 glands on the lower lid during 10-15 seconds. Total of 15 glands are evaluated along the lower eyelid margin, consisting of five glands located in each of the temporal, central, and nasal regions. For each of the 15 glands, expressed secretion characteristics were graded as 3 (clear liquid secretion), 2 (cloudy liquid secretion), 1 (inspissated/toothpaste consistency), and 0 (no secretion). This is the Meibomian Gland Score (MGS).
  For data analysis, the MGS score for each eye was calculated based on the sum of the secretion grades for all 15 glands evaluated with a range of 0 to 45. Lower score means a better function of meibomian glands.

CONTACTS AND LOCATIONS:
Overall Officials: Margarita Calonge Cano, MD, PhD, Principal Investigator — Study Principal Investigator
Locations (1):
- Instituto Universitario de Oftalmobiología Aplicada (IOBA), Valladolid, Spain

IPD SHARING:
Plan to Share IPD: No